CLINICAL TRIAL: NCT03810157
Title: Does Laser-assisted Hatching(LAH) May Improve the Pregnancy Outcomes in Human?
Brief Title: Does LAH May Improve the Pregnancy Outcomes?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1215
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Pregnancy Outcomes
Keywords: laser-assisted hatching (LAH); zona pellucida; cryopreservation; pregnancy outcomes

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser-assisted hatching system (Experimental): Embryos were exposed to a dose of laser energy focused outside the zona pellucida by aser-assisted hatching system.
  Interventions: Device: Laser-assisted hatching system
- Control group (No Intervention): Nothing is done.

INTERVENTIONS:
Device: Laser-assisted hatching system — The ZP was thinned or drilled with the Laser-assisted hatching system. The laser pulse was 0.296 ms. Laser aperture was 8μm.
  Arms: Laser-assisted hatching system

SUMMARY:
A defect in the hatching stage is considered an important cause of implantation failure. Therefore, assisted hatching (AH), which involves artificial disruption of the zona pellucida, has been proposed as a method for improving the capacity of the embryo to implant. But the advantage of using laser to facilitate the hatching process of embryos in ART practice is debatable, and an optimum strategy for performing LAH remains elusive. Therefore, the aim of this study was to evaluate the effects of laser-assisted hatching(LAH) on clinical outcomes. Patients were randomly divided into control and LAH groups. The zona pellucida was thinned or drilled with a diode laser. Relevant parameters are recorded to evaluate the validity of LAH in ART.

DETAILED DESCRIPTION:
Hatching is a very important process for successful implantation involving the breaking of the embryo out of the zona pellucida at the blastocyst stage. Inadequate hatching of the blastocyst might lead to implantation failure in ART. Currently, a variety of AH techniques have been used including zona thinning and the opening or complete removal of the zona by laser. But the advantage of using laser to facilitate the hatching process of embryos in ART practice is debatable, and an optimum strategy for performing LAH remains elusive. Therefore, the investigator aim to discuss the effectiveness of LAH in ART.

In this study, patients were randomly divided into control and LAH groups. A quarter of zona pellucida of the cleavage-stage embryo was thinned to 6.6 μm. All operation was performed in the empty region without contact to the blastomere in order to minimize the blastomere damage. The ZP of blastocyst was drilled with laser, the ZP opening 20% of its initial length. The operation was performed in the opposite region of ICM in order to minimize the damage. In the control group, embryos were transplanted without LAH. The rate of clinical pregnancy, live-birth, miscarriage, multiple gestation were evaluated. This research intends to discuss whether LAH can improve the clinical outcomes in ART, and further choice the appropriate LAH action site.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF/ICSI-ET cycle；
* The zone pellucida of the cleavage-stage embryo is thicker than 8 μm.

Exclusion Criteria:

* Number of embryos transferred per cycle >2;
* The transferred embryos including fresh and frozen cycle in the same cycle;
* Embryos developed from the frozen-thawed oocytes.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2018-12-26 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of LAH in ART | 6 months
  Assess the clinical pregnancy

SECONDARY OUTCOMES:
Feasibility of LAH in ART | 1 year
  Incidence of LAH adverse events was assessed by miscarriage rate and multiple gestation rate.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Li, Study Chair — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China